CLINICAL TRIAL: NCT06879054
Title: Lifestyle, Education, Activity, Nutrition (LEAN) Into Pregnancy: A Randomized Controlled Trial Investigating the Impact of Healthy Lifestyle Education During Preconception and Early Pregnancy on Cardiovascular and Pregnancy Outcomes
Brief Title: Lifestyle, Education, Activity, Nutrition (LEAN) Into Pregnancy
Acronym: LEAN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Anna Palatnik, MD, Associate Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO48098
Record Dates: First submitted 2025-02-14; First posted 2025-03-17 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Pregnancy; Preconception Education; Preconception Care, Preconception Risk; Adverse Pregnancy Outcomes
Keywords: Preconception education; Cardiovascular health; Pregnancy; Lifestyle intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LEAN Intervention (Experimental): Participants randomized to the LEAN Intervention arm will complete five modules on nutrition for optimal health and submit their completed certificates. The Gaples Institute is a free website that provides free educational modules regarding nutrition education. Each module is 10-15 minutes long and covers the power of a healthy diet, the truth about dietary fat, information about carbohydrates, facts about protein, calcium, and sodium, and simple strategies for healthy eating. Participants will also receive weekly phone calls to follow up with the progress of the implementation of the lifestyle intervention for the next three months.
  Interventions: Other: Healthy lifestyle education
- Standard of Care (No Intervention): Participants randomized to the Standard of Care arm will receive routine prenatal or gynecologic care.

INTERVENTIONS:
Other: Healthy lifestyle education — Healthy lifestyle education via nutritional educational modules from the Gaples Institute.
  Other Names: Health lifestyle education
  Arms: LEAN Intervention

SUMMARY:
The goal of this randomized controlled clinical trial is to determine if healthy lifestyle education can help improve cardiovascular health and reduce pregnancy complications in women during the preconception period or early pregnancy. The main aims include:

1. Determine the feasibility and acceptability of the LEAN into pregnancy study.
2. Determine the impact of healthy lifestyle education on Life's Essential 8 cardiovascular health score.
3. Determine the impact of health lifestyle education on adverse pregnancy outcomes, specifically gestational diabetes and preeclampsia.

A total of 200 participants will be randomly assigned to receive healthy lifestyle education in addition to routine care, or routine care alone. Participants will be asked to participate in the following activities:

* Blood draws to test hemoglobin A1c and lipids
* Surveys about diet, physical activity, sleep, and tobacco use
* Gaples Nutritional Education Modules (if applicable)

DETAILED DESCRIPTION:
Studies investigating adverse pregnancy outcomes have shown contributing effects from increased rates of diabetes, hypertension, and abnormal cholesterol and cardiovascular disease events. Previous studies have additionally shown that lifestyle modifications such as the DASH diet, regular exercise, and reduction in stress can lower blood pressure, lower LDL cholesterol levels, and decrease poor health behaviors that are linked to cardiovascular disease. However, studies have failed to quantify the effects of lifestyle modifications on more short-term cardiovascular health that may increase adverse pregnancy outcomes. By shifting the focus from cardiovascular disease treatment to positive health promotion, it promotes a paradigm shift to focus on prevention of disease and improved societal health overall. Preliminary data from our group showed significant correlations between preeclampsia and lower availability of healthy food, which is one of the factors quantified in Life's Essential 8. A major gap in the literature remains lifestyle interventions that can lead to risk factors for cardiovascular health in pregnant populations during gestation and also in the preconception period. We believe that lifestyle interventions preconception or during pregnancy can improve cardiovascular health during gestation and reduce adverse pregnancy outcomes.

We hypothesize that the implementation of specific educational modules surrounding diet and exercise and repeated patient interaction will improve Life's Essential 8 cardiovascular score and, in those who are pregnant, potentially reduce the risk for gestational diabetes and preeclampsia.

ELIGIBILITY:
Inclusion Criteria:

* Patients in a period of preconception who want to become pregnant within 2 years, or patients in their first trimester of pregnancy
* English-speaking
* At risk for preeclampsia based on the following ACOG criteria: ≥1 high-risk factor: history of preeclampsia, multifetal gestation, chronic hypertension, gestational hypertension, pregestational diabetes, renal disease, or autoimmune disease, OR ≥2 moderate-risk factors: nulliparity, obesity (BMI>30 kg/m2), family history of preeclampsia, Black or African American race, age ≥35 years, or personal history factors (previous pregnancy low birth weight, previous stillbirth, previous preterm birth, >10-year pregnancy interval).
* At risk for gestational diabetes, defined by ACOG as a BMI > 25 plus one or more of the following risk factors: physical inactivity, first-degree relative with diabetes, high-risk race/ethnicity (African American, Latino, Native American, Asian American, Pacific Islander), previous infant weight >4,000g, previous GDM, chronic hypertension, HDL <35, triglyceride >250, PCOS, A1c ≥ 5.7, prepregnancy BMI >40.

Exclusion Criteria:

* No access to a smartphone
* Major fetal anomaly diagnosed during current pregnancy, if pregnant at consent

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2029-05 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the LEAN into Pregnancy Study | From enrollment through the end of intervention at 3 months.
  Determine feasibility (as measured by recruitment, completion of all modules and surveys, and retention in the study for three months) of the LEAN into Pregnancy study.

SECONDARY OUTCOMES:
Life's Essential 8 | At enrollment and after intervention at 3 months.
  Determine the impact of healthy lifestyle education on Life's Essential 8 cardiovascular score pre- and post-intervention.
Incident rate of gestational diabetes among participants who become pregnant. | Up to 2 years after enrollment
  Determine the impact of healthy lifestyle education on adverse pregnancy outcomes among participants who become pregnant, specifically the rate of gestational diabetes.
Acceptability of the LEAN into Pregnancy Study | 3 months from enrollment (end of intervention)
  Acceptability will be measured by surveys distributed to participants in the intervention arm at the final study visit.
Incident rate of hypertensive disorders of pregnancy in participants who become pregnant | Up to 2 years after enrollment
  Determine the impact of healthy lifestyle education on adverse pregnancy outcomes among participants who become pregnant, specifically the rate of hypertensive disorders of pregnancy.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Palatnik, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No